CLINICAL TRIAL: NCT02965053
Title: A Single-center, Randomized, 2-Period, Crossover, Study to Explore The Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of EOS789 in Patients With Chronic Kidney Disease and Hyperphosphatemia on Hemodialysis
Brief Title: A Phase1 Study to Explore the Safety of EOS789 in Patients With Chronic Kidney Disease and Hyperphosphatemia on Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EOS103US
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Period 1 Arm 1 (Experimental): EOS789 Dose 1 in treatment sequence 1, Placebo in treatment sequence 2
  Interventions: Drug: EOS789; Drug: Placebo
- Period 1 Arm 2 (Experimental): Placebo in treatment sequence 1, EOS789 Dose 1 in treatment sequence 2
  Interventions: Drug: EOS789; Drug: Placebo
- Period 2 Arm 1 (Experimental): EOS789 Dose 2 in treatment sequence 1, EOS789 Dose 2 + Sevelamer carbonate in treatment sequence 2
  Interventions: Drug: EOS789; Drug: Renvela
- Period 2 Arm 2 (Experimental): EOS789 Dose 2 + Sevelamer carbonate in treatment sequence 1, EOS789 Dose 2 in treatment sequence 2
  Interventions: Drug: EOS789; Drug: Renvela

INTERVENTIONS:
Drug: EOS789
Drug: Placebo
  Arms: Period 1 Arm 1; Period 1 Arm 2
Drug: Renvela
  Other Names: Sevelamer carbonate
  Arms: Period 2 Arm 1; Period 2 Arm 2

SUMMARY:
This study is a randomized study designed as a 2x2 cross-over in two periods (Period 1 and Period 2) to assess the safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of EOS789 in patients with chronic kidney disease (CKD) and hyperphosphatemia receiving hemodialysis. Period 1 is double-blind and Period 2 is open-label. Period 1 and Period 2 are identical with regard to the design, inclusion/exclusion criteria, and assessments. EOS789 and its combination with sevelamer carbonate are tested in Period 1 and Period 2 respectively.

ELIGIBILITY:
Inclusion Criteria:

- Patients with CKD and hyperphosphatemia must meet the following criteria for study entry:

* Age ≥18 years
* On thrice-weekly hemodialysis for at least 3 months prior to screening
* Not having changed dialysis prescription within 4 weeks prior to screening for dialyzer, calcium concentration in dialysate, or dry weight more than 1 kg
* Receiving stable doses of treatments affecting serum phosphorus for at least 4 weeks prior to screening and willing to discontinue these treatments

Exclusion Criteria:

- Patients with CKD and hyperphosphatemia who meet any of the following criteria will be excluded from study entry:

* Uncontrolled diabetes and/or hypertension in the opinion of the investigators
* Uncontrolled chronic constipation and/or diarrhea in the opinion of the investigators
* Hospitalization for cardiac disease in previous 3 months
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Safety: Incidences of adverse events | Up to Day 42 in each treatment sequence
  Incidences of adverse events
Safety: Change from baseline in vital signs | Up to Day 42 in each treatment sequence
  Change from baseline in vital signs (systolic blood pressure, diastolic blood pressure, pulse rate)
Safety: Change from baseline in clinical laboratory tests | Up to Day 42 in each treatment sequence
  Change from baseline in clinical laboratory tests (hematology, biochemistry, coagulation)
Safety: Change from baseline in 12 lead ECGs | Up to Day 42 in each treatment sequence
  Change from baseline in 12 lead ECGs

SECONDARY OUTCOMES:
Pharmacokinetics: Plasma concentration of EOS789 | Day 4, 9, 10, 11 in the first treatment sequence in each period
Pharmacokinetics: Total exposure (area under the curve [AUC]) | Day 10 in the first treatment sequence in each period
Pharmacokinetics: Maximum concentration (Cmax) | Day 10 in the first treatment sequence in each period
Pharmacokinetics: Time to reach Cmax (Tmax) | Day 10 in the first treatment sequence in each period
Pharmacokinetics: Removal ratio of EOS789 by hemodialysis at steady state | Day 9 in the first treatment sequence in each period
Pharmacodynamics: Intestinal fractional phosphorus absorption and accumulated fecal excretion of phosphorus | Days 11 to 13 in the first treatment sequence and second treatment sequence in each period
Efficacy: Change from baseline of serum phosphorus (P), Calcium (Ca), Ca x P, intact parathyroid hormone (PTH), and fibroblast growth factor (FGF23) at Day 13 | Day 13 in the first treatment sequence and second treatment sequence in each period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Leader, Study Director — Chugai Pharmaceutical
Locations (1):
- Indianapolis, Indiana, United States